CLINICAL TRIAL: NCT01634867
Title: A Pilot Study of Intubating Conditions Comparing Intraosseous Vascular Access With Peripheral Intravenous Access for Drug Delivery in Rapid Sequence Intubation Using Rocuronium as the Paralytic Agent
Brief Title: Observational Study of Rapid Sequence Intubation (RSI) Drug Delivery Using Intraosseous (IO) and Intravenous (IV) Access in Pediatric Patients
Status: Withdrawn | Type: Observational
Why Stopped: No subject enrollment.
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-03
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Airway Control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intraosseous (IO) drug delivery: patients in whom intraosseous (IO) vascular access has been established for rapid sequence intubation drug delivery.
- Peripheral intravenous (IV) drug delivery: patients in whom peripheral intravenous (IV) vascular access has been established for rapid sequence intubation drug delivery.

SUMMARY:
This study will evaluate using intraosseous vascular access and intravenous vascular access to give pediatric patients the necessary medications to perform rapid sequence intubation, for patients with airway difficulties.

ELIGIBILITY:
Inclusion Criteria:

* subjects requiring rapid sequence intubation for whom rocuronium is chosen as the paralytic agent.
* the operator chooses to place a peripheral intravenous or powered intraosseous catheter to permit rapid sequence intubation.

Exclusion Criteria:

* subjects in whom vascular access for rapid sequence intubation drug administration was established prior to arrival to the emergency department.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients in the emergency department with airway difficulties requiring rapid sequence intubation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Time from determination of need for vascular access for rapid sequence intubation to administration of first does of paralytic agent. | during rapid sequence intubation procedure, average expected time frame 30 minutes
Time from vascular access to intubation first attempt, as indicated by the first attempt to visualize the larynx with the laryngoscope. | during rapid sequence intubation procedure, average expected time frame 30 minutes
time from vascular access to successful intubation | during rapid sequence intubation procedure, average expected time frame 30 minutes
number of attempts necessary for successful intubation | during rapid sequence intubation procedure, average expected time frame 30 minutes

SECONDARY OUTCOMES:
Intubation difficulty | during rapid sequence intubation procedure, average time frame 30 minutes
  The Intubation Difficulty Scale is a validated tool used to grade the difficulty with which a patient was intubated for airway managment during rapid sequence intubation.
operator satisfaction with intubating conditions | during rapid sequence intubation procedure, average time frame 30 minutes
failure rate of endotracheal intubation | during rapid sequence intubation procedure, average time frame 30 minutes
  failure rate of endotracheal intubation and requirement for alternative airway management.
Time from presentation of patient to vascular access established | during rapid sequence intubation procedure, average time frame 30 minutes
Determine the incidence of short term catheter related complications for each technique | during emergency department stay, average time frame 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Edward Truemper, MD, Principal Investigator — University of Nebraska
Locations (1):
- Omaha Children's Hospital and Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Reades R, Studnek JR, Vandeventer S, Garrett J. Intraosseous versus intravenous vascular access during out-of-hospital cardiac arrest: a randomized controlled trial. Ann Emerg Med. 2011 Dec;58(6):509-16. doi: 10.1016/j.annemergmed.2011.07.020. PMID 21856044
- [Background] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Background] Leidel BA, Kirchhoff C, Bogner V, Braunstein V, Biberthaler P, Kanz KG. Comparison of intraosseous versus central venous vascular access in adults under resuscitation in the emergency department with inaccessible peripheral veins. Resuscitation. 2012 Jan;83(1):40-5. doi: 10.1016/j.resuscitation.2011.08.017. Epub 2011 Sep 3. PMID 21893125
- [Background] Deakin CD, Nolan JP, Soar J, Sunde K, Koster RW, Smith GB, Perkins GD. European Resuscitation Council Guidelines for Resuscitation 2010 Section 4. Adult advanced life support. Resuscitation. 2010 Oct;81(10):1305-52. doi: 10.1016/j.resuscitation.2010.08.017. No abstract available. PMID 20956049
- [Background] Kleinman ME, de Caen AR, Chameides L, Atkins DL, Berg RA, Berg MD, Bhanji F, Biarent D, Bingham R, Coovadia AH, Hazinski MF, Hickey RW, Nadkarni VM, Reis AG, Rodriguez-Nunez A, Tibballs J, Zaritsky AL, Zideman D; Pediatric Basic and Advanced Life Support Chapter Collaborators. Part 10: Pediatric basic and advanced life support: 2010 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2010 Oct 19;122(16 Suppl 2):S466-515. doi: 10.1161/CIRCULATIONAHA.110.971093. PMID 20956258
- [Background] Brierley J, Carcillo JA, Choong K, Cornell T, Decaen A, Deymann A, Doctor A, Davis A, Duff J, Dugas MA, Duncan A, Evans B, Feldman J, Felmet K, Fisher G, Frankel L, Jeffries H, Greenwald B, Gutierrez J, Hall M, Han YY, Hanson J, Hazelzet J, Hernan L, Kiff J, Kissoon N, Kon A, Irazuzta J, Lin J, Lorts A, Mariscalco M, Mehta R, Nadel S, Nguyen T, Nicholson C, Peters M, Okhuysen-Cawley R, Poulton T, Relves M, Rodriguez A, Rozenfeld R, Schnitzler E, Shanley T, Kache S, Skippen P, Torres A, von Dessauer B, Weingarten J, Yeh T, Zaritsky A, Stojadinovic B, Zimmerman J, Zuckerberg A. Clinical practice parameters for hemodynamic support of pediatric and neonatal septic shock: 2007 update from the American College of Critical Care Medicine. Crit Care Med. 2009 Feb;37(2):666-88. doi: 10.1097/CCM.0b013e31819323c6. PMID 19325359
- [Background] Von Hoff DD, Kuhn JG, Burris HA 3rd, Miller LJ. Does intraosseous equal intravenous? A pharmacokinetic study. Am J Emerg Med. 2008 Jan;26(1):31-8. doi: 10.1016/j.ajem.2007.03.024. PMID 18082778
- [Background] Orlowski JP, Porembka DT, Gallagher JM, Lockrem JD, VanLente F. Comparison study of intraosseous, central intravenous, and peripheral intravenous infusions of emergency drugs. Am J Dis Child. 1990 Jan;144(1):112-7. doi: 10.1001/archpedi.1990.02150250124049. PMID 1688484
- [Background] Laurin EG, Sakles JC, Panacek EA, Rantapaa AA, Redd J. A comparison of succinylcholine and rocuronium for rapid-sequence intubation of emergency department patients. Acad Emerg Med. 2000 Dec;7(12):1362-9. doi: 10.1111/j.1553-2712.2000.tb00493.x. PMID 11099426
- [Background] Perry JJ, Lee JS, Sillberg VA, Wells GA. Rocuronium versus succinylcholine for rapid sequence induction intubation. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD002788. doi: 10.1002/14651858.CD002788.pub2. PMID 18425883